CLINICAL TRIAL: NCT05577767
Title: Does Longitudinal Nursing Follow-up Improve Smoking Cessation in Patients With Chronic Obstructive Pulmonary Disease (COPD) Screening
Brief Title: Does Longitudinal Nursing Follow-up Improve Smoking Cessation in Patients Referred for COPD Screening
Acronym: BPCO
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier de Valence (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH-CHV-02
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: COPD; Nurse's Role
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
a monocentric study to evaluate the efficacy of a longitudinal nursing follow up in smoking cessation in patients screened for Chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
The challenges to limit the occurrence of COPD are early detection, the fight against smoking and smoking and addictions (e.g. Cannabis), as well as the fight against environmental exposures.

we proposed to evaluate if a longitudinal nursing follow-up at 3 months, 6 months and one year, in patients coming to screening for COPD.

Cessation of respiratory toxics is the most effective intervention in stopping the progression of COPD.

ELIGIBILITY:
Inclusion Criteria:

* Smoking patients screened for COPD between 35 years old 65 years old
* Read, write and understand the French language
* Patient affiliated to a social security system
* Written and signed informed consent

Exclusion Criteria:

* Patients with a diagnosis of respiratory diseases
* Patients receiving inhaled respiratory therapy
* Persons unable to perform spirometry
* Pregnant women
* Refusal to participate in research
* Patient under guardianship, deprived of liberty, safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Smoking patients screened for COPD between 35 years old 65 years old
Sampling Method: Non-Probability Sample
Enrollment: 233 (Estimated)
Dates: Start 2020-09-11 (Actual); Primary Completion 2025-09-11 (Estimated); Study Completion 2026-09-11 (Estimated)

PRIMARY OUTCOMES:
number of cigarettes or other toxic substances | up to 1 year
  per day

CONTACTS AND LOCATIONS:
Overall Officials: Gilles RIVAL, MD, Principal Investigator — CH VALENCE
Locations (1):
- Ch Valence, Valence, Drome, France

IPD SHARING:
Plan to Share IPD: Undecided